



# **Statistical Analysis Plan**

Version 2.0, February 2025

NCT06191848

### **Authors:**

Dr Sharmala Thuraisingam A/Prof Tim Spelman Dr Cade Shadbolt A/Prof Chris Schilling Prof Michelle Dowsey

## **Table of Contents**

| 1. Adı | ministrative Information | 5 |
|---------|-----------------------------------------------------|----|
| 1.1 | L Study identifiers | 5 |
| 1.2 | 2 Revision history | 5 |
| 1.3 | Contributors to the statistical analysis plan | 5 |
| 1.4 | 4 Approvals | 5 |
| 2. Intr | roduction | 5 |
| 3. Stu | udy synopsis | 6 |
| 4. Stu | udy objectives | 6 |
| 4.1 | l Primary objective | 6 |
| 4.2 | 2 Secondary objective | 6 |
| 4.3 | 3 Safety objective | 6 |
| 5. Pat | tient population | 6 |
| 5.1 | I Inclusion criteria | 6 |
| 5.2 | 2 Exclusion criteria | 7 |
| 6. Stu | udy outcomes | 7 |
| 6.1 | L Primary outcome | 7 |
| 6.2 | 2 Secondary outcomes | 7 |
| 6.3 | 3 Safety outcomes | 8 |
| 7. Inte | ervention | 9 |
| 8. Rar | ndomisation and blinding | 9 |
| 9. Sar | mple size | 10 |
| 10. St | tatistical analysis | 10 |
| 10. | .1 General principles | 10 |
| 10. | .2 Interim analyses | 10 |
| 10. | .3 Multiplicity adjustment | 10 |
| 10. | .4 Data sets to be analysed | 10 |
| 10. | .5 Participant disposition | 11 |
| 10. | .6 Patient characteristics and baseline comparisons | 11 |
| 10. | .7 Analysis of the primary outcome | 11 |
| | 10.7.1 Main analysis | |

| 10.7.2 Sensitivity analyses | 11 |
|-----------------------------------------|----|
| 10.7.3 Subgroup analyses | 11 |
| 10.8 Analysis of secondary outcomes | 12 |
| 10.8.1 Continuous secondary outcomes | 12 |
| 10.8.2 Binary secondary outcomes | 12 |
| 10.8.3 Time to event secondary outcomes | 12 |
| 10.9 Treatment of missing data | 12 |
| 10.10 Health economic assessment | 12 |
| 10.11 Analysis of safety outcomes | 13 |
| 11. References | 14 |
| Appendix 1: Proposed tables and figures | 16 |

### **List of Abbreviations**

AE Adverse event

AOANJRR Australian Orthopaedic Association National Joint Replacement Registry

BMI Body Mass Index
CI Confidence interval

FDA Food and Drug Administration

ICH International Council for Harmonisation

IQR Interquartile range

IPTW Inverse Probability of Treatment Weighting

ITT Intention to treat

MCS Mental component score
NDI National Death Index

OA Osteoarthritis

PASE Physical activity scale for the elderly

PCS Physical component score

RR Relative risk

SAE Serious adverse event SAP Statistical analysis plan

SF Short Form

SHR Subdistribution hazard ratio

VDI Victorian Death Index

WOMAC Western Ontario and McMaster Universities Arthritis Index

## 1. Administrative Information

This statistical analysis plan is based on the study protocol version 2.0 dated 28th November 2024.

### 1.1 Study identifiers

ClinicalTrials.gov register NCT06191848.

### 1.2 Revision history

| Version | Date | Changes made to document | Authors |
|---|---|---|---|
| 1.0 | 06/12/2024 | First draft | Sharmala Thuraisingam |
| 2.0 | 28/02/2025 | Revised following initial feedback | Sharmala Thuraisingam |

### 1.3 Contributors to the statistical analysis plan

| Names and ORCID | Affiliation | Role on study | SAP contribution |
|---|---|---|---|
| Dr Sharmala Thuraisingam<br>0000-0002-9450-1302 | University of Melbourne,<br>Department of Surgery, St<br>Vincent's Hospital | Statistician | Statistical concepts and writing of plan |
| A/Prof Tim Spelman<br>0000-0001-9204-3216 | University of Melbourne,<br>Department of Surgery, St<br>Vincent's Hospital | Senior Statistician | Statistical concepts and writing of plan |
| Dr Cade Shadbolt<br>0000-0002-0937-2412 | University of Melbourne,<br>Department of Surgery, St<br>Vincent's Hospital | Data Scientist | Statistical concepts and contributions to plan |
| A/Prof Chris Schilling<br>0000-0002-1747-7249 | University of Melbourne,<br>Department of Surgery, St<br>Vincent's Hospital | Health Economist | Health economic concepts and writing of plan |
| Prof Michelle Dowsey<br>0000-0002-9708-5308 | University of Melbourne,<br>Department of Surgery, St<br>Vincent's Hospital | Principal Investigator | Statistical concepts and contributions to plan |

### 1.4 Approvals

All authors have reviewed this plan and approve it as final. They find it to be consistent with the requirements of the protocol as it applies to their respective areas. They also find it to be compliant with ICH-E9 principles and, in particular, confirm that this analysis plan was developed in a completely blinded manner (i.e. without knowledge of the effect of the intervention(s) being assessed).

### 2. Introduction

This statistical analysis plan (SAP) details the intended analyses to be conducted on data collected in the STOP KNEE-OA trial. The SAP includes the primary and secondary analyses, health economic assessments, as well as the proposed layout

of tables and figures for the main outcome paper. All analyses detailed in this plan have been pre-specified prior to the completion of data collection and comply with the FDA's Guidance for Industry ICH E9 Statistical Principles for Clinical Trials.

## 3. Study synopsis

STOP KNEE-OA is a multicentre, double-blinded, parallel group, randomised controlled trial designed to determine if weekly subcutaneous tirzepatide is superior to placebo in limiting the progression to knee replacement in adults with moderate-to-severe knee osteoarthritis who were eligible for unilateral knee replacement, with a body-mass index (BMI) of at least 30 kg/m², without diabetes. Participants will be randomised in a 1:1 ratio to the tirzepatide and placebo study arms, and all participants will receive standardised dietary and physical activity advice. Follow-up of participants will occur every 4 weeks for 72 weeks through on-site and telephone visits. Long term follow-up at 5 and 10 years will be achieved through data linkage with the Australian Orthopaedic Association National Joint Replacement Registry (AOANJRR) and the National Death Index (NDI)/Victorian Death Index (VDI) (1,2).

### 4. Study objectives

### 4.1 Primary objective

The primary efficacy aim is to determine whether weekly tirzepatide added to standardised lifestyle advice compared with standardised lifestyle advice only (placebo), reduces the proportion of participants that progress to knee replacement surgery within 72 weeks. The primary null hypothesis of no difference in the proportion of participants that progress to knee replacement in participants assigned to tirzepatide versus placebo within 72 weeks will be tested.

### 4.2 Secondary objective

The secondary efficacy aims are to evaluate whether weekly tirzepatide is superior to placebo in: (1) improving osteoarthritis symptoms, (2) reducing patient's willingness to undergo knee replacement, (3) reducing bodyweight, (4) improving physical and mental health status, (5) improving physical activity levels, (6) reducing the use of prescription pain medication at 72 weeks and (7) reducing the proportion of patients that progress to knee replacement within 5 and 10 years. In each case, the null hypothesis of no difference between study arms will be tested.

### 4.3 Safety objective

The safety aims are to determine whether weekly tirzepatide are associated with adverse events, serious adverse events and adverse events that require treatment discontinuation.

## 5. Patient population

#### 5.1 Inclusion criteria

Participants will be eligible to participate in the trial if they provide informed consent and meet all the following criteria:

- Age ≥ 18 years
- BMI ≥30 kg/m<sup>2</sup>

- Been unsuccessful in losing body weight through lifestyle modification.
- Deemed eligible by an orthopaedic surgeon to be on the waiting list at one of the participating sites for primary knee replacement surgery in the target joint due to osteoarthritis.
- Moderate-to-severe osteoarthritis in the target joint as defined by Kellgren-Lawrence grade ≥2.
- Willing to and capable of self-injecting tirzepatide and following study procedures for the duration of the trial.
- Female participants must not be pregnant, breastfeeding nor of reproductive potential (further details in study protocol)

#### 5.2 Exclusion criteria

Participants will be ineligible to participate in the trial if they meet any of the following criteria:

- Deemed eligible by an orthopaedic surgeon to be on the waiting list at one of the participating sites for knee replacement surgery in the contralateral knee.
- Used prescription medication for weight loss in the three months prior to screening.
- Undergone surgical or endoscopic procedures for weight loss in the past.
- Diagnosed with type 1 or 2 diabetes.
- Have laboratory evidence of diabetes mellitus during screening.
- Have a personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN 2).
- Have an active malignancy excluding basal or squamous cell skin cancer.
- Awaiting or have a transplanted organ.
- Have received chronic systemic glucocorticoid therapy (for more than 14 days) in prior 3 months or have a significant, active autoimmune abnormality (e.g., lupus or rheumatoid arthritis) that the study doctor deems likely to require systemic glucocorticoid therapy during the next 18 months.
- Have any other medical condition, abnormal laboratory tests or medications as outlined in the protocol section 5.3.2 that makes them unsuitable to participate in the trial.
- Are part of the study site team/personnel or family member of the study site team/personnel.
- Currently enrolled in any other study of an investigational product or previously enrolled in another study within 90 days of study visit 1.

### 6. Study outcomes

### **6.1 Primary outcome**

The primary outcome is the proportion of patients that progress to knee replacement surgery at 72 weeks. The effect estimate is the relative risk of knee replacement surgery at 72 weeks (tirzepatide vs placebo).

### **6.2 Secondary outcomes**

Secondary outcomes for the main analysis and health economic assessment are summarised in Table 1.

## **6.3 Safety outcomes**

Safety outcomes have been defined in the study protocol and include adverse events (AE), serious adverse events (SAE) and adverse events requiring treatment discontinuation that occur any time throughout the 72-week trial period.

| Table 1. Secondary o | utcome measu | res | | | |
|---|---|---|---|---|---|
| Main Analysis | Variable | Effect estimates | Assessment time | Analysis set | Statistical |
| · | type | | points | | model |
| Change in WOMAC pain | Continuous | Mean difference in change in WOMAC pain | 72 weeks | FAS | Linear<br>mixed<br>model |
| Change in WOMAC function | Continuous | Mean difference in change in WOMAC function | 72 weeks | FAS | Linear<br>mixed<br>model |
| Change in WOMAC stiffness | Continuous | Mean difference in change in WOMAC stiffness | 72 weeks | FAS | Linear<br>mixed<br>model |
| Willingness for surgery* | Binary | Relative risk | 72 weeks | FAS | Binomial regression |
| Percentage change in body weight | Continuous | Mean difference in percentage change in body weight | 72 weeks | FAS | Linear<br>mixed<br>model |
| ≥5% reduction in body weight | Binary | Relative risk | 72 weeks | FAS | Binomial regression |
| ≥10% reduction in body weight | Binary | Relative risk | 72 weeks | FAS | Binomial regression |
| ≥20% reduction in bodyweight | Binary | Relative risk | 72 weeks | FAS | Binomial regression |
| Change in SF-36<br>MCS | Continuous | Mean difference in change in SF-36 MCS | 72 weeks | FAS | Linear<br>mixed<br>model |
| Change in SF-36 PCS | Continuous | Mean difference in change in SF-36 PCS | 72 weeks | FAS | Linear<br>mixed<br>model |
| Change in PASE | Continuous | Mean difference in change in PASE | 72 weeks | FAS | Linear<br>mixed<br>model |
| Use of non-opioid prescription analgesics | Binary | Relative risk | 68-72 weeks | FAS | Binomial regression |
| Use of opioid prescription analgesics | Binary | Relative risk | 68-72 weeks | FAS | Binomial regression |
| Opioid prescription analgesic dose | Continuous | Mean difference in oral<br>morphine equivalent (OME)<br>per day (3) | 72 weeks | FAS | Linear<br>mixed<br>model |
| Knee replacement surgery (long term) | Time to event with death as | Subdistribution hazard ratio | 5 and 10 years | FAS | Fine & Gray<br>competing<br>risk model |

| | competing risk | | | | |
|---|---|---|---|---|---|
| Health Economic Analysis | | | | | |
| Change in health-<br>related quality of<br>life using SF-36 | Continuous | Mean difference in Quality<br>Adjusted Life Years (QALY) | 3 monthly until 72<br>weeks, 5 and 10<br>years | FAS | Linear and<br>generalized<br>linear<br>models |
| Cost-effectiveness | Ratio | Incremental cost-<br>effectiveness ratio (cost per<br>QALY) | 72 weeks, 5 and<br>10 years | FAS | Linear and<br>generalized<br>linear<br>models |

<sup>\*</sup>Patients will be considered willing to undergo surgery at 72 weeks if they had a knee replacement by 72 weeks or remained on the surgery waiting list.

Abbreviations: WOMAC=Western Ontario and McMaster Universities Osteoarthritis Index; MCS=mental component score; PCS=Physical Component Score; PASE=Physical Activity Scale for the Elderly; SF-36=36-Item Short Form Health Survey; QALY=Quality-adjusted life-year; FAS=Full Analysis Set.

#### 7. Intervention

Participants will be randomised to receive either tirzepatide or placebo and self-administer the pre-filled syringes subcutaneously into the thigh or abdomen on a weekly basis for 72 weeks. Administration of the drug/placebo will occur on the same day, at approximately the same time, each week. Intervention participants will initially receive 2.5mg of tirzepatide which will be increased by 2.5mg every four weeks over the 20-week dose escalation period until the target weekly dose of 15mg is reached. Participants who are unable to reach the target weekly dose will remain at the highest tolerable dose of either 5mg or 10mg. Dose modifications will only be permitted for participants experiencing gastrointestinal symptoms and will be addressed as outlined in the protocol (section 5.5.3 Dose escalation and modification). Participants that require their dose of tirzepatide reduced below 5mg will discontinue the study drug.

All participants will receive dietary and physical activity counselling throughout the study, including advice on making healthy food choices and achieving calculated calorie deficits.

## 8. Randomisation and blinding

Randomisation of participants will occur at the second study visit, after participant screening and consent have occurred. The study's Interactive Web Response Systems (IWRS) will randomly allocate participants to either the tirzepatide or placebo group in a 1:1 ratio using randomly permuted block sizes of 2 and 4. Randomisation will be stratified by site, gender (male or female) and body mass index (BMI) category (30-39.9 kg/m² or 40+ kg/m²).

All investigators, site personnel and statisticians will be blinded to participant study group allocations. Only the study pharmacist at the central pharmacy will be unblinded to ensure the correct medication and dosages are dispensed to participants. Individual site pharmacists will remain blinded.

## 9. Sample size

To detect a 10% reduction in progression to knee replacement surgery at 72 weeks from 95% in the placebo group to 85% in the tirzepatide group (with 80% power, two-tailed  $\alpha$ =0.05), and 10% attrition rate, a sample size of 352 participants (176 per group) is required. The sample size is based on the ABS Study (4), a randomized controlled trial that demonstrated a 24.4% (95% CI 9.0% to 39.8%) reduction in progression to knee replacement surgery in surgical weight loss (gastric banding) participants compared with participants who received lifestyle modification advice. The effect size for the sample size calculation is based on the lower limit of the 95% confidence interval for the effect size observed in the ABS study. The estimated attrition rate of 10% and assumed 95% progression to knee replacement in the placebo arm is based on the ABS study and other trials investigating the progression to orthopaedic surgery ((4–6). The sample size calculation was performed in Stata version 18 (StataCorp. 2023. Stata Statistical Software: Release 18. College Station, TX: StataCorp LLC.) using the "sampsi" command, which allows for continuity correction (7).

## 10. Statistical analysis

### 10.1 General principles

The following sections provide further detail on the primary and secondary analyses stated in the study protocol.

All data cleaning and statistical analyses will be conducted using Stata version 18 (StataCorp. 2023. Stata Statistical Software: Release 18. College Station, TX: StataCorp LLC.)(7). Statistical tests will be two-tailed and a p-value<0.05 used to determine statistical significance. Continuous data will be summarised using means, standard deviations (SD) and range, and medians and interquartile ranges (IQR) for skewed data. Categorical data will be summarised using counts and percentages. Transformations will be tested when modelling skewed continuous outcomes. Results from analyses will be accompanied by 95% confidence intervals and p-values.

### 10.2 Interim analyses

No interim analyses for efficacy, futility and/or sample size revision are pre-planned for this trial. The Data Monitoring Committee may request and conduct unplanned interim analyses if required.

### 10.3 Multiplicity adjustment

No formal adjustments for multiplicity are planned given there is only one primary outcome. However, the multiple comparisons, strength of evidence and consistency of effects across the outcomes will be considered when interpreting the secondary analyses results.

### 10.4 Data sets to be analysed

All primary and secondary analyses will be performed using the full analysis set. This data set will include all data obtained from all participants randomised in the trial regardless of whether they adhered to or discontinued the study drug. Outcome data for knee replacement at 72 weeks will be obtained through data linkage with the Australian Orthopaedic Association National Joint Replacement Registry (AOANJRR) (1). To facilitate the analysis of long-term outcomes, knee replacement data (from AOANJRR) will be linked at 5 and 10 years, along with dates of death from the National Death Index (NDI)/Victorian Death Index (VDI) (2). The safety analysis data set will include all participants randomised in the trial and any adverse event data.

#### 10.5 Participant disposition

A CONSORT flowchart (Appendix 1, Figure 1) will be prepared to summarise the number of participants who were screened for eligibility, excluded, randomised and withdrew. Reasons for exclusion and withdrawal will be listed.

### 10.6 Patient characteristics and baseline comparisons

Participant characteristics at baseline will be summarised by trial arm and presented as outlined in Appendix 1 Table 1. Descriptive statistics will be used to compare baseline characteristics between the study arms.

#### 10.7 Analysis of the primary outcome

#### 10.7.1 Main analysis

The "treatment-regimen" estimand (8) will compare the proportion of participants in each of the assigned treatment groups that progress to knee replacement within 72-weeks regardless of adherence to study drug. Binomial regression will be used to estimate the relative risk of knee replacement at 72 weeks in the intervention arm compared with the placebo arm. Results will be presented as shown in Appendix 1 Table 4. Point estimate relative risks and risk differences will be presented with associated 95% confidence intervals. A graph depicting the cumulative incidence of knee replacement with time will be presented (Appendix 1, Figure 5).

#### 10.7.2 Sensitivity analyses

Three sensitivity analyses will be conducted on the primary outcome:

- (1) An adjusted analysis which extends the main analysis model to include stratification variables. Two different models will be fit. The first will include site, gender and BMI as fixed effects, the second model will include these stratification variables as random effects.
- (2) Time to knee replacement will be analysed using a Cox proportional hazards model with treatment included as a covariate. The treatment effect will be estimated by the hazard ratio (HR) and 95% confidence interval.
- (3) The "trial product" estimand (hypothetical strategy) (8) provides an estimate of the treatment effect had participants remained on their treatment for the planned 72-week treatment duration. The estimand is based on a hypothetical scenario in which intercurrent events do not occur (8). In this study, intercurrent events are defined as discontinuation of treatment due to adverse events or for other reasons outlined in the protocol (8). Either mixed models or Inverse Probability of Treatment Weighting (IPTW) with or without multiple imputation may be used for the "trial product" estimand (9,10).

Treatment effect estimates obtained from the sensitivity analyses will be included in a forest plot (Appendix 1, Figure 6) alongside the "treatment-regimen" estimand.

#### 10.7.3 Subgroup analyses

The primary analysis as defined in section 10.7.1, will be conducted according to the following subgroups defined by baseline characteristics:

- 1. Sex (male, female)
- 2. Body Mass Index (30 to 40, ≥40 kg/m<sup>2</sup>)
- 3. Kellgren-Lawrence Grade (2, 3 or 4)

For each subgroup analysis, the subgroup variable and an interaction between subgroup and treatment will be included as fixed effects in the model. The significance of the interaction term (P<0.05) will be used to assess whether treatment effects differ across the levels of the subgroup. Treatment effect estimates from the subgroup analyses will be included in a forest plot with estimates from the main and sensitivity analyses (Appendix 1, Figure 6).

### 10.8 Analysis of secondary outcomes

The "treatment-regimen" estimand (8) will be estimated for all secondary outcomes. Where mixed models are used, random intercepts will be included to account for clustering of the outcome within participants and an unstructured variance-covariance structure assumed. Treatment effect estimates will be adjusted by stratification factors. Appendix 1, Tables 5-7 show the intended table layouts for the results, and Figures 7-13 the planned plots.

#### 10.8.1 Continuous secondary outcomes

For the continuous secondary outcomes listed in Table 1, linear mixed models using restricted maximum likelihood estimation will be used to estimate the difference in mean outcome between the arms at 72 weeks. The outcome at 3-monthly intervals will be included as dependent variables in the model. The outcome at baseline, time and an interaction between time and treatment group will be included as fixed effects in the model.

#### 10.8.2 Binary secondary outcomes

Binomial regression models will be used to estimate the relative risk of willingness for surgery, reduction in body weight ( $\geq$ 5%,  $\geq$ 10% and  $\geq$ 20%) and use of opioid and non-opioid prescription analgesics (Table 1) in the tirzepatide arm compared with the placebo arm at 72 weeks.

#### 10.8.3 Time to event secondary outcomes

Fine & Gray competing risk regression models will be used to estimate the rate of knee replacement (subdistribution hazard rate) in the tirzepatide arm compared with the placebo arm at 5 and 10 years. Death will be treated as a competing risk given the age of the study population.

### 10.9 Treatment of missing data

It is anticipated that there will not be any missing outcome data for the primary outcome given the occurrence of knee replacement at 72 weeks will be determined through in person study visits, review of hospital records and linkage with the Australian Orthopaedic Association National Joint Replacement Registry (AOANJRR) which has near complete capture of all knee replacements in Australia (1). However, should data linkage be delayed, and/or there be less than 40% missing outcome data, multiple imputation may be used, subject to approval by the Data Safety Monitoring Board. Imputation models will include the outcome, stratification factors and any auxiliary variables available in the data set that may explain the missing outcome data. The validity of the imputed data will be assessed via graphical comparisons of imputed and observed data, including kernel density plots and histograms, and comparisons of goodness-of-fit between imputed and non-imputed datasets. The same approach will be used for secondary outcomes where there are less than 40% missing data.

#### 10.10 Health economic assessment

A cost-utility analysis will be completed to assess the cost-effectiveness of treatment relative to the status quo standardised lifestyle advice. First, the trial results will be considered without any further extrapolation. Outcomes will be Quality Adjusted Life Years (QALYs), calculated via linear interpolation of health-related quality of life measures from

the SF-36 at baseline and each follow-up measurement. A health system perspective will be adopted, with costs including the intervention and follow-up treatment, in particular joint replacement. A cost-effectiveness plane and cost-acceptability curve will be presented. A subsequent step may also be included, extrapolating the results of the longer-term impact of the trial results for a further 5 and 10 years using the Australian Osteoarthritis (AUS-OA) validated health economic model (12), using a discount rate of 3.5%. A probabilistic sensitivity analysis would be incorporated to assess the robustness of the model-based results to changes in the input parameters and assumptions. Results will be presented as shown in Appendix 1, Table 8 and Figures 14-15.

### 10.11 Analysis of safety outcomes

For each event type (AE and SAE), the number and proportion of participants experiencing the event, median number of events and rate of events will be reported by study group. The proportion of participants that experience a fatal event or an adverse event resulting in treatment discontinuation will also be reported. Adverse events occurring in over 5% of participants in any of the trial arms will be summarised. Results will be presented as shown in Appendix 1, Table 9.

### 11. References

- 1. South Australian Health and Medical Research Institute. Home AOANJRR [Internet]. 2019 [cited 2020 Apr 24]. Available from: https://aoanjrr.sahmri.com/
- 2. Australian Institute of Health and Welfare. National Death Index (NDI) Australian Institute of Health and Welfare [Internet]. 2020 [cited 2020 Apr 24]. Available from: https://www.aihw.gov.au/about-our-data/our-data-collections/national-death-index
- 3. Nielsen S, Degenhardt L, Hoban B, Gisev N. A synthesis of oral morphine equivalents (OME) for opioid utilisation studies. Pharmacoepidemiol Drug Saf [Internet]. 2016 Jun 1 [cited 2024 Dec 3];25(6):733–7. Available from: https://onlinelibrary.wiley.com/doi/full/10.1002/pds.3945
- 4. Dowsey MM, Brown WA, Cochrane A, Burton PR, Liew D, Choong PF. Effect of Bariatric Surgery on Risk of Complications After Total Knee Arthroplasty: A Randomized Clinical Trial. JAMA Netw Open [Internet]. 2022 Apr 1 [cited 2024 Jul 10];5(4):e226722–e226722. Available from: https://jamanetwork.com/journals/jamanetworkopen/fullarticle/2791035
- 5. Dowsey MM, Gould DJ, Spelman T, Pandy MG, Choong PF. A Randomized Controlled Trial Comparing a Medial Stabilized Total Knee Prosthesis to a Cruciate Retaining and Posterior Stabilized Design: A Report of the Clinical and Functional Outcomes Following Total Knee Replacement. J Arthroplasty [Internet]. 2020 Jun 1 [cited 2024 Jul 10];35(6):1583-1590.e2. Available from: https://pubmed.ncbi.nlm.nih.gov/32139194/
- 6. Dowsey M, Castle D, Knowles S, Monshat K, Salzberg M, Nelson E, et al. The effect of mindfulness training prior to total joint arthroplasty on post-operative pain and physical function: A randomised controlled trial. Complement Ther Med [Internet]. 2019 Oct 1 [cited 2024 Jul 10];46:195–201. Available from: https://pubmed.ncbi.nlm.nih.gov/31519279/
- 7. StataCorp LLC. Stata | Data Analysis and Statistical Software [Internet]. 2018 [cited 2018 Mar 12]. Available from: https://www.stata.com/products/
- 8. European Medicines Agency Committee for Medicinal Products for Human Use. ICH E9 (R1) addendum on estimands and sensitivity analysis in clinical trials to the guideline on statistical principles for clinical trials. 2020 [cited 2024 Sep 23]; Available from: https://www.ema.europa.eu/en/documents/scientific-guideline/ich-e9-r1-addendum-estimands-and-sensitivity-analysis-clinical-trials-guideline-statistical-principles-clinical-trials-step-5\_en.pdf
- 9. Jastreboff AM, Aronne LJ, Ahmad NN, Wharton S, Connery L, Alves B, et al. Tirzepatide Once Weekly for the Treatment of Obesity. New England Journal of Medicine [Internet]. 2022 Jul 21 [cited 2024 Dec 3];387(3):205–16. Available from: https://www.nejm.org/doi/full/10.1056/NEJMoa2206038
- 10. Parra CO, Daniel RM, Wright D, Bartlett JW. Estimating hypothetical estimands with causal inference and missing data estimators in a diabetes trial. 2023 Aug 24 [cited 2024 Dec 6]; Available from: https://arxiv.org/abs/2308.13085v2
- 11. Bond S, Allison A. rpsftm: rank-preserving structural failure time models for survival data. 2024.

15

Schilling C, Zhou Y, Rele S, Shadbolt C, Thuraisingam S, O'Brien P, et al. The development of AUS-OA - a population

12.

## **Appendix 1: Proposed tables and figures**

Figure 1: Consort flowchart



Figure 2a: Data linkage reporting flowchart at 72 weeks



Figure 2b: Data linkage reporting flowchart at 5 and 10 years



**Table 1:** Baseline characteristics

| | Total (N=) | Tirzepatide (N=) | Placebo (N=) |
|-------------------|------------|------------------|--------------|
| | n (%) | n (%) | n (%) |
| Demographics | | | |
| Age, median [IQR] | | | |
| Female | | | |
| etc. | | | |
| Clinical measures | | | |
| BMI (kg/m²) | | | |
| 30-39.9 | | | |
| ≥40 | | | |
| etc. | | | |
| Sites | | | |
| etc. | | | |

Figure 3. Dosing of tirzepatide and placebo over trial period

Table 2: Reasons for discontinuing allocated treatment by study group

Figure 4. Cumulative proportion of patients who discontinued treatment by study group

Table 3: Concomitant therapies by study group

 Table 4: Analysis of primary outcome (treatment-regimen estimand)

| | Tirzepatide<br>(N=) | Placebo<br>(N=) | Unadjusted | | | |
|---|---|---|---|---|---|---|
| | n (%) | n (%) | RR (95% CI) | P-value | RD (95% CI) | P-value |
| Knee | | | | | | |
| replacement | | | | | | |
| at 72 weeks | | | | | | |

Abbreviations: RR= relative risk, RD=risk difference, CI=confidence interval

Figure 5. Cumulative incidence (%) of knee replacement with time

Figure 6. Forest plot of treatment effect estimates at 72 weeks from primary, sensitivity and subgroup analyses

Table 5: Analysis of continuous secondary outcomes (treatment-regimen estimand)

| | Tirzepatide (N=) | | Placebo (N=) | | Adjusted | |
|---|---|---|---|---|---|---|
| | N | Estimated mean<br>(95% CI) | N | Estimated mean<br>(95% CI) | Tirzepatide vs<br>placebo between-<br>group differences<br>(95% CI) | P-value |
| Change in WOMAC pain at 72 weeks | | | | | | |

| Change in WOMAC function at 72 weeks |
|----------------------------------------------------|
| Change in WOMAC stiffness at 72 weeks |
| Percentage change<br>in body weight at 72<br>weeks |
| Change in SF-36<br>MCS at 72 weeks |
| Change in SF-36 PCS at 72 weeks |
| Change in PASE at 72 weeks |
| OME per day at 68-<br>72 weeks |

Note: All change estimates are from baseline.

Abbreviations: CI=confidence interval, WOMAC=Western Ontario and McMaster Universities Arthritis Index, SF-36=36-Item short form survey, PCS=physical component summary, MCS=mental component summary, PASE=physical activity scale for the elderly, OME=oral morphine equivalent.

Figures 7-13: Graphs for longitudinal secondary outcomes (WOMAC pain, WOMAC function, WOMAC stiffness, body weight, SF-36 MCS, SF-36 PCS, PASE) (a) effect estimates at 3-monthly time intervals and (b) cumulative frequency of change from baseline.

**Table 6:** Analysis of binary secondary outcomes

| | Tirzepatide<br>(N=) | Placebo<br>(N=) | Adjusted | | | |
|---|---|---|---|---|---|---|
| | n (%) | n (%) | RR (95% CI) | P-value | RD (95% CI) | P-value |
| ≥5% reduction in body | | | | | | |
| weight at 72 weeks | | | | | | |
| ≥10% reduction in | | | | | | |
| body weight at 72 | | | | | | |
| weeks | | | | | | |
| ≥20% reduction in | | | | | | |
| body weight at 72 | | | | | | |
| weeks | | | | | | |
| Willingness for surgery | | | | | | |
| at 72 weeks | | | | | | |
| Use of non-opioid | | | | | | |
| prescription analgesics | | | | | | |
| at 68-72 weeks | | | | | | |
| Use of opioid | | | | | | _ |
| prescription analgesics | | | | | | |
| at 68-72 weeks | | | | | | |

Abbreviations: RR=relative risk, RD=risk difference, CI=confidence interval

**Table 7.** Analysis of secondary time to event outcomes

| | Tirzepatide (N=) | Placebo (N=) | Adjusted | |
|------------------|------------------|--------------|--------------|---------|
| Knee replacement | n (%) | n (%) | SHR (95% CI) | P-value |
| 5 years | | | | |
| 10 years | | | | |

Abbreviations: SHR=subdistribution hazard ratio, CI=confidence interval

**Table 8:** Health economics analysis

| | Tirzepatide (N=) | Placebo (N=) | Difference |
|---|---|---|---|
| QALYs | | | |
| Costs | | | |
| Incremental cost effectiveness ratio (ICER) | | | |

Abbreviations: QALYs = Quality Adjusted Life Years

Figure 14: Cost-effectiveness plane

Figure 15: Cost acceptability curve

**Table 9: Adverse drug events** 

| | Total (N=) | Tirzepatide (N=) | Placebo (N=) |
|---|---|---|---|
| Any adverse event | | | |
| At least one adverse event, n(%) | | | |
| Median number of adverse events, median [IQR] | | | |
| Rate of adverse events, (events per person) | | | |
| Event type | | | |
| Adverse event (AE) | | | |
| At least one, n(%) | | | |
| Median number, median [IQR] | | | |
| Rate, (events per person) | | | |
| Serious adverse event (SAE) | | | |
| At least, n(%) | | | |
| Median number, median [IQR] | | | |
| Rate, (events per person) | | | |
| Adverse event requiring treatment discontinuation, n(%) | | | |
| Fatal event, n(%) | | | |
| Specific adverse events reported in more than 5% of | | | |
| participants in any group, n(%) | | | |

Abbreviations: AE=adverse event, SAE=serious adverse event